CLINICAL TRIAL: NCT00142051
Title: Inhaled Nitric Oxide for Pediatric Painful Sickle Crisis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 18 or 20 enrolled, stopped due to paucity of available participants
Sponsor: Boston Children's Hospital (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Debra Weiner, Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-09-119; FD-R-002560-01 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; pain crisis; vaso-occlusive crisis; nitric oxide
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Nitric Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): inhaled NO
  Interventions: Drug: nitric oxide
- 2 (Placebo Comparator): room air inhalation
  Interventions: Drug: oxygen

INTERVENTIONS:
Drug: nitric oxide — 80 ppm 8 hrs, 40 ppm 8 hrs, 20 ppm 4 hrs, 10 ppm 4 hrs
  Arms: 1
Drug: oxygen — oxygen fi02 21% (room air)
  Arms: 2

SUMMARY:
Randomized, double blind placebo controlled clinical trial to evaluate effectiveness and safety of inhaled nitric oxide for the treatment of sickle cell painful crisis in pediatric patients with sickle cell disease.

DETAILED DESCRIPTION:
The specific aim of this study is to evaluate the clinical effectiveness of inhaled nitric oxide (INO) for the treatment of acute vaso-occlusive pain crisis in pediatric patients with sickle cell disease. Nitric oxide (NO) deficiency is known to be central to the pathophysiology of vaso-occlusion. The aim is unchanged from the original application. The study is a randomized, double blind, placebo controlled, clinical trial with eligible patients randomized to receive either NO (with 21% O2 final concentration) for 16 hrs with 8 hr wean (80 ppm 0-8 hrs, 40 ppm 9-16 hrs, 20 ppm 17-20 hrs, 10 ppm 21-24 hrs) or placebo (21% O2 alone) for 24 hrs. The null hypothesis is that there is no difference in change in mean pain score after 16 hours between patients treated with NO and placebo. The primary outcome measure of the study remains the difference in mean change in pain scores between groups as assessed using a 10 cm visual analogue pain scale (VAS). Secondary outcome measures also remain the same. The study is a next step to our completed FDA Orphan Product Development Grant funded study (FD-R-001686) that evaluated safety and efficacy of NO used for 4 hrs for treatment of vaso-occlusive crisis in pediatric patients with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

1. Hemoglobin SS, Hemoglobin Sß0thal or Hemoglobin SC documented by prior hemoglobin electrophoresis.
2. Age 9 years or greater, age 22 years or less; pediatric age range, old enough to comply with mask and give reliable pain assessment score.
3. Acute pain crisis defined as pain in abdomen, back and/or extremities that cannot be explained by a diagnosis other than sickle cell disease.
4. Initial pain score at least 6 cm; to optimize the likelihood of observing a significant difference in change in pain score between INO treated and placebo groups. Based on data from our previous study, it is anticipated that patients will have an average pre-inhalation pain score of approximately 8 cm.

Exclusion Criteria:

1. > 24 pain crises in the last 12 months. Patients with very frequent pain crisis may have biologic and/or psychosocial pathophysiology that differs from those with fewer pain crises.
2. Pain crisis treated at a medical facility within the last 12 hours.
3. Use of investigational drugs other than hydroxyurea within the last 30 days.
4. Significant respiratory compromise (initial SaO2 < 90%) and/or patients likely to have acute chest syndrome (chest pain and infiltrate) will be eliminated.
5. Clinically significant acute or chronic cardiac dysfunction.
6. Acute priapism.
7. New focal neurologic symptoms.
8. Concurrent documented or suspected bacterial or parvovirus infection.
9. Temperature > 38.4ºC. These patients may have concomitant infection.
10. Transfusion within 30 days or chronic transfusion therapy.
11. Pregnant female
12. Cigarette smoker > 1/2 ppd.
13. Allergy to morphine

    -

Ages: 9 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2005-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Difference in change in mean pain score (visual analog scale) after 16 hours of treatment between patients treated with INO and placebo. | every 4 hrs x duration of hospitalization

SECONDARY OUTCOMES:
Secondary outcome measures to evaluate efficacy | Duration of hospitalization, followup
Longitudinal analyses of change in VAS pain score over 16 hours. | every 4 hrs, duration of hospitalization
Change in pain score using a 5 point descriptive scale and a 5 point relief scale. | every 4 hours duration of hospitalization
Time to pain score less than 5 cm for 2 consecutive VAS pain assessments 4 hours apart and not using parenteral narcotics. | every 4 hrs, duration of hospitalization
Use of pain medication: cumulative dose of parenteral narcotic pain medications. | While patient on parenteral narcotic
Duration of hospitalization. | Time of discharge
Inflammatory markers/mediators. | 0, 16 and q 24 hrs during hospitalization
Secondary outcome measures to evaluate safety are: | 4, 8, 16, 24 hrs methb, constant NO2, 02 during inhalation
Maximum concentration of methemoglobin. | 0, 4, 8, 16, 24 hrs
Maximum concentration of nitrogen dioxide (NO2) delivered. | continuous over 24 hrs of inhalaiton
Minimum percent oxygen saturation of hemoglobin (by pulse oximetry). | continuous over 24 hrs of inhalation then every 4 hrs for duration of hospitalization
Maximum and minimum vital signs: pulse, respiratory rate, blood pressure. | every 4 hrs during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Debra Weiner, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gladwin MT, Kato GJ, Weiner D, Onyekwere OC, Dampier C, Hsu L, Hagar RW, Howard T, Nuss R, Okam MM, Tremonti CK, Berman B, Villella A, Krishnamurti L, Lanzkron S, Castro O, Gordeuk VR, Coles WA, Peters-Lawrence M, Nichols J, Hall MK, Hildesheim M, Blackwelder WC, Baldassarre J, Casella JF; DeNOVO Investigators. Nitric oxide for inhalation in the acute treatment of sickle cell pain crisis: a randomized controlled trial. JAMA. 2011 Mar 2;305(9):893-902. doi: 10.1001/jama.2011.235. PMID 21364138
- [Background] Weiner DL, Hibberd PL, Betit P, Cooper AB, Botelho CA, Brugnara C. Preliminary assessment of inhaled nitric oxide for acute vaso-occlusive crisis in pediatric patients with sickle cell disease. JAMA. 2003 Mar 5;289(9):1136-42. doi: 10.1001/jama.289.9.1136. PMID 12622584